CLINICAL TRIAL: NCT06105034
Title: Placenta Accreta Spectrum Disorder Conservative Managment Versus Hysterectomy Prospective Analysis
Status: Completed | Type: Observational
Sponsor: Nourhan Elsadany (Other)
Responsible Party: Sponsor-Investigator, Nourhan Elsadany, sponsor investigator, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: MS 714/2021
Record Dates: First submitted 2022-05-11; First posted 2023-10-27 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Placenta Accreta
Keywords: placenta accreta spectrum managment
MeSH Terms: conditions — Placenta Accreta | interventions — Suture Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conservative management: 150 patients
  Interventions: Procedure: interventional techniques, the severity of placental invasion, and various placental positions and suture techniques
- CS hysterectomy: 150 patients
  Interventions: Procedure: interventional techniques, the severity of placental invasion, and various placental positions and suture techniques

INTERVENTIONS:
Procedure: interventional techniques, the severity of placental invasion, and various placental positions and suture techniques — Clinically, severe complications of PA include severe obstetric hemorrhage leading to disseminated intravascular coagulopathy (DIC), iatrogenic injury to the ureters, bladder, bowel, respiratory distress syndrome (RDS), acute transfusion reactions, electrolyte imbalance, and renal failure. In women with PA, the expected blood loss at delivery is 3000- 5000 mL, About 90% of patients require a blood transfusion with 40% requiring more than ten units of packed cell transfusion

SUMMARY:
The aim of this study is to identify risk factors associated with performing cesarean hysterectomy versus conservative management in patients with placenta accreta spectrum (PAS).

Research question What are the risk factors associated with cesarean hysterectomy in patients with placenta accreta spectrum? Research hypothesis There are certain risk factors associated with cesarean hysterectomy in patients with Placenta accreta spectrum (PAS).

DETAILED DESCRIPTION:
Placenta accreta spectrum disorder (PAS) is a serious obstetric disorder that is characterized by low lying and deep penetration of the villi which are abnormally attached to the myometrium of the uterus. This obstructs its complete separation during the third stage of labor which induces continued bleeding, and have potentially life- threatening for the mother. Most commonly, it is a consequence of a partial or complete absence of the compact and spongy layer known as the decidua basalis, and mis-development of the fibrinoid Nitabuch's layer which lies between the boundary zone of the thick endometrium and the cytotrophoblastic shell in the placenta.

Traditionally, caesarean hysterectomy at the time of delivery has been the preferred management strategy for placenta previa accreta. Not only does this approach preclude future fertility, but it is also a procedure synonymous with signiﬁcant perioperative risks. For women who wish to conserve their reproductive function, other treatment options have been described.

1.INTRODUCTION/ REVIEW Placenta accreta is defined as "the abnormal localization and adherence of the placenta villi to the uterine myometrium. Patients at risk for abnormal placentation should be assessed antenally by ultrasonography, with or without adjunct magnetic resonance imaging if indicated . Various grading systems of villous invasion during placenta implantation are integrated to a spectrum (PAS), including placenta accreta (the villi invade superficially into the myometrium), increta (the villi invade deeper into the myometrium but do not reach the serosa), and percreta (the villi invade into the uterine serosa or adjacent organs) Clinically, severe complications of PA include severe obstetric hemorrhage leading to disseminated intravascular coagulopathy (DIC), iatrogenic injury to the ureters, bladder, bowel, respiratory distress syndrome (RDS), acute transfusion reactions, electrolyte imbalance, and renal failure. In women with PA, the expected blood loss at delivery is 3000- 5000 mL, About 90% of patients require a blood transfusion with 40% requiring more than ten units of packed cell transfusion .

The most difficult problem to deal with is controlling hemorrhage during delivery caused by PAS disorders. The potential for bleeding correlates with the degree to which the placenta invades the myometrium, the area of abnormal adherence involved, and the presence or absence of invasion into extrauterine tissues such as the bladder or parametrial tissues .

Different methods have been employed to manage the PA, ranging from uterine conservation, which involves leaving the placenta in situ, to conventional hysterectomy. Classical cesarean sections (C- sections) prevent the excessive bleeding by leaving the adherent placenta in situ and by adopting strategic planning with a comprehensive analysis that aids the reduction in maternal morbidity and mortality rates .

Perinatal emergency hysterectomy is routinely used to avoid maternal morbidity and mortality . Given the fact that cesarean section history and placenta previa are major risk factors, the incidence of PAS disorders increases with the increasing rate of cesarean section .

Other risk factors include spontaneous or induced abortion, repeated miscarriages, in vitro fertilization embryo transfer, advanced maternal age, history of endometrial ablation, and previous uterine surgery .

Conservative and non-conservative management for PAS disorders have been compared. Cesarean hysterectomy is regarded as the safest and most practical, thereby remaining the management option of choice. Nevertheless, hysterectomy is associated with high rates of severe maternal morbidity. In cases of placenta percreta, especially with bladder invasion, owing to damage to pelvic organs and vasculature during hysterectomy .In recent years, with the application of an abdominal artery balloon and the improvement of surgical techniques, efforts are made to preserve the uterus for patients PAS. This is not only the improvement for fertility preservation, but also for better control of bleeding to reduce maternal morbidity.

The evidence on conservative management is considered low-quality, less reproducible, and operator-dependent. Critics noted the lack of histopathological confirmation or detailed differential diagnosis. Confounding factors in these studies needs to be controlled including the application of interventional techniques, the severity of placental invasion, and various placental positions and suture techniques .

Therefore, investigators will undertake a prospective study to analyze maternal and neonatal outcomes comparing women with PAS disorders treated with cesarean hysterectomy or conservatively.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with history of previous cesarean section.
* Age above 18 years.
* Gestational age above 28 weeks.
* Confirmed diagnosis of Placenta previa accreta spectrum disorder by U/S or MRI if needed.
* U/S signs suggestive of placenta previa accrete (Green-top Guideline).

Exclusion Criteria:

* Gestational age less than 28 weeks.
* Age less than 18years

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The aim of this study is to identify risk factors associated with performing cesarean hysterectomy versus conservative management in patients with placenta accreta spectrum (PAS).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Number of the patient who diagnosed intraoperative with placenta accreta spectrum disorder and undergoing conservative management or hysterectomy | from time of operation to diagnoses 1week
  The diagnoses will be made based on intra-operative findings and/or pathologic features depending on the degree of placenta invasion (invading the myometrium or invading up to or beyond the uterine serosa). Patients with placenta accreta with complete peri-operative information will be included for further analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Nourhan Abdelhady Soliman Elsadany, Giza, Egypt

REFERENCES:
- [Background] Zeng C, Yang M, Ding Y, Duan S, Zhou Y. Placenta accreta spectrum disorder trends in the context of the universal two-child policy in China and the risk of hysterectomy. Int J Gynaecol Obstet. 2018 Mar;140(3):312-318. doi: 10.1002/ijgo.12418. Epub 2018 Jan 16. PMID 29214633
- [Background] Yan J, Shi CY, Yu L, Yang HX. Folding Sutures Following Tourniquet Binding as a Conservative Surgical Approach for Placenta Previa Combined with Morbidly Adherent Placenta. Chin Med J (Engl). 2015 Oct 20;128(20):2818-20. doi: 10.4103/0366-6999.167365. No abstract available. PMID 26481753
- [Background] Wang Q, Ma J, Zhang H, Dou R, Huang B, Wang X, Zhao X, Chen D, Ding Y, Ding H, Cui S, Zhang W, Xin H, Gu W, Hu Y, Ding G, Qi H, Fan L, Ma Y, Lu J, Yang Y, Lin L, Luo X, Zhang X, Fan S, Yang H. Conservative management versus cesarean hysterectomy in patients with placenta increta or percreta. J Matern Fetal Neonatal Med. 2022 May;35(10):1944-1950. doi: 10.1080/14767058.2020.1774871. Epub 2020 Jun 4. PMID 32498575
- [Background] Thurn L, Lindqvist PG, Jakobsson M, Colmorn LB, Klungsoyr K, Bjarnadottir RI, Tapper AM, Bordahl PE, Gottvall K, Petersen KB, Krebs L, Gissler M, Langhoff-Roos J, Kallen K. Abnormally invasive placenta-prevalence, risk factors and antenatal suspicion: results from a large population-based pregnancy cohort study in the Nordic countries. BJOG. 2016 Jul;123(8):1348-55. doi: 10.1111/1471-0528.13547. Epub 2015 Jul 29. PMID 26227006
- [Background] Silver RM, Fox KA, Barton JR, Abuhamad AZ, Simhan H, Huls CK, Belfort MA, Wright JD. Center of excellence for placenta accreta. Am J Obstet Gynecol. 2015 May;212(5):561-8. doi: 10.1016/j.ajog.2014.11.018. Epub 2014 Nov 20. PMID 25460838
- [Background] Silver RM. Abnormal Placentation: Placenta Previa, Vasa Previa, and Placenta Accreta. Obstet Gynecol. 2015 Sep;126(3):654-668. doi: 10.1097/AOG.0000000000001005. PMID 26244528
- [Background] Sentilhes L, Kayem G, Chandraharan E, Palacios-Jaraquemada J, Jauniaux E; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Conservative management. Int J Gynaecol Obstet. 2018 Mar;140(3):291-298. doi: 10.1002/ijgo.12410. No abstract available. PMID 29405320
- [Background] Sentilhes L, Goffinet F, Kayem G. Management of placenta accreta. Acta Obstet Gynecol Scand. 2013 Oct;92(10):1125-34. doi: 10.1111/aogs.12222. PMID 23869630
- [Background] Sentilhes L, Ambroselli C, Kayem G, Provansal M, Fernandez H, Perrotin F, Winer N, Pierre F, Benachi A, Dreyfus M, Bauville E, Mahieu-Caputo D, Marpeau L, Descamps P, Goffinet F, Bretelle F. Maternal outcome after conservative treatment of placenta accreta. Obstet Gynecol. 2010 Mar;115(3):526-534. doi: 10.1097/AOG.0b013e3181d066d4. PMID 20177283
- [Background] Liu HY, Lin XG, Wu JL, Qiao FY, Deng DR, Zeng WJ. [Multiposition spiral suture of the lower uterine segment: a new technique to control the intraoperative bleeding of pernicious placenta previa]. Zhonghua Fu Chan Ke Za Zhi. 2016 Oct 25;51(10):754-758. doi: 10.3760/cma.j.issn.0529-567X.2016.10.009. Chinese. PMID 27788743
- [Background] Licon E, Matsuzaki S, Opara KN, Machida H, Roman LD, Sasso EB, Matsuo K. Treatment and outcome of placenta percreta: Primary cesarean hysterectomy versus conservative management. Eur J Obstet Gynecol Reprod Biol. 2020 Jan;244:201-203. doi: 10.1016/j.ejogrb.2019.09.017. Epub 2019 Sep 20. No abstract available. PMID 31627939
- [Background] Latif Khan Y, Rahim A, Gardezi J, Iqbal M, Hassan Z, Altaf S, Bhatti S. Conventional and conservative management of placenta accreta is two ends of a single continuum: A report of three cases and literature review. Clin Case Rep. 2018 Jul 13;6(9):1739-1746. doi: 10.1002/ccr3.1717. eCollection 2018 Sep. PMID 30214754
- [Background] Jauniaux E, Alfirevic Z, Bhide AG, Belfort MA, Burton GJ, Collins SL, Dornan S, Jurkovic D, Kayem G, Kingdom J, Silver R, Sentilhes L; Royal College of Obstetricians and Gynaecologists. Placenta Praevia and Placenta Accreta: Diagnosis and Management: Green-top Guideline No. 27a. BJOG. 2019 Jan;126(1):e1-e48. doi: 10.1111/1471-0528.15306. Epub 2018 Sep 27. No abstract available. PMID 30260097
- [Background] Hunt JC. Conservative management of placenta accreta in a multiparous woman. J Pregnancy. 2010;2010:329618. doi: 10.1155/2010/329618. Epub 2010 Sep 30. PMID 21490740
- [Background] Society of Gynecologic Oncology; American College of Obstetricians and Gynecologists and the Society for Maternal-Fetal Medicine; Cahill AG, Beigi R, Heine RP, Silver RM, Wax JR. Placenta Accreta Spectrum. Am J Obstet Gynecol. 2018 Dec;219(6):B2-B16. doi: 10.1016/j.ajog.2018.09.042. PMID 30471891
- [Background] Bowman ZS, Eller AG, Bardsley TR, Greene T, Varner MW, Silver RM. Risk factors for placenta accreta: a large prospective cohort. Am J Perinatol. 2014 Oct;31(9):799-804. doi: 10.1055/s-0033-1361833. Epub 2013 Dec 12. PMID 24338130
- [Result] Zhao X, Tao Y, Du Y, Zhao L, Liu C, Zhou Y, Wei P. The application of uterine wall local resection and reconstruction to preserve the uterus for the management of morbidly adherent placenta: Case series. Taiwan J Obstet Gynecol. 2018 Apr;57(2):276-282. doi: 10.1016/j.tjog.2018.02.017. PMID 29673673